CLINICAL TRIAL: NCT02422576
Title: Efficacy of Natural Ingredient to Improve the Swallowing Response of Patients With Oropharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14.13.NRC
Record Dates: First submitted 2015-03-24; First posted 2015-04-21 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — lemon balm leaf extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control + Product 1 (Active Comparator): Control product (Thicken Up clear: TUC) + natural ingredient 1 (cinnamon extract)
  Interventions: Other: cinnamon extract; Other: Thicken Up clear: TUC
- Control + Product 2 (Active Comparator): Control product (Thicken Up clear: TUC) + natural ingredient 2 (lemon extract)
  Interventions: Other: lemon extract; Other: Thicken Up clear: TUC
- Control + Product 3 (Active Comparator): Control product (Thicken Up clear: TUC) + natural ingredient 3 (lemon extract+eucalyptus extract)
  Interventions: Other: lemon extract plus eucalyptus extract; Other: Thicken Up clear: TUC

INTERVENTIONS:
Other: cinnamon extract — acute exposure to natural ingredient during physiological parameters recording (deglutition or cortical activity)
  Arms: Control + Product 1
Other: lemon extract — acute exposure to natural ingredient during physiological parameters recording (deglutition or cortical activity)
  Arms: Control + Product 2
Other: lemon extract plus eucalyptus extract — acute exposure to natural ingredient during physiological parameters recording (deglutition or cortical activity)
  Arms: Control + Product 3
Other: Thicken Up clear: TUC

SUMMARY:
Assessment of the improvement of the safety of the swallowing function under 3 natural ingredients known to be agonist of sensory receptors.

DETAILED DESCRIPTION:
The trial will be double-blind, randomized, monocentric, and interventional with a hybrid design. The subjects will be randomized to one of the three parallel active ingredient groups. Products will be compared versus control (Thicken Up Clear - nectar viscosity), which adds a part of cross over within the design.

The total sample size is 84 enrolled subjects. Patients will be males and females aged 55+ with mild proven dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 55+
* Patients showing impaired safety of the deglutition during the V-VST (volume - viscosity swallow test): Cough oxygen desaturation ≥3% or voice change.
* Neurodegenerative or ischemic/hemorrhagic cerebral cause (stroke) or elderly subjects

Exclusion Criteria:

* Patients radiated for treatment of head and neck cancer Idiosyncrasis
* Allergy to food or medication, especially contrast products (iodine)
* Major respiratory disease needing oxygen as standard treatment.
* Any major and relevant abdominal, head and neck, or chest surgery within the three months preceding the study.
* Have a high alcohol consumption (more than 2 drinks/day)
* Subject who cannot be expected to comply with the study procedures, including consuming the test products.
* Currently participating or having participated in another clinical trial during the month preceding the study
* Patients with relevant mucosal damage or with in-mouth irritation
* Patients with pacemaker or electrode implants
* Epileptic patients

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06-12 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Improvement of the safety of the swallowing function, according to Rosenbek's scale | up to15 min after ingredient ingestion
  The maximum PAS score across the different boluses (5, 10 and 20 ml) during nectar series (with and without active ingredient) assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.

SECONDARY OUTCOMES:
Swallowing safety-Prevalence of penetration | up to15 min after ingredient ingestion
  the prevalence of penetration in the population according to Rosenbek's PAS (scores of 2-5)
  , assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Swallowing safety-Prevalence of aspiration | up to15 min after ingredient ingestion
  the prevalence of aspiration in the population according to Rosenbek's PAS (scores of 6-8), assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Efficacy of swallowing function-Severity of the amount of oral and pharyngeal residues | up to15 min after ingredient ingestion
  Severity of the amount of oral and pharyngeal residues, assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Efficacy of swallowing function-Prevalence of subjects with oral and pharyngeal residues | up to15 min after ingredient ingestion
  Prevalence of subjects with oral and pharyngeal residues, assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Efficacy of swallowing function-Time to upper oesophageal sphincter opening | up to15 min after ingredient ingestion
  Time to upper oesophageal sphincter opening, assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Efficacy of swallowing function-Time to laryngeal vestibule opening | up to15 min after ingredient ingestion
  Time to laryngeal vestibule opening, assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Efficacy of swallowing function-time to laryngeal vestibule closure | up to15 min after ingredient ingestion
  time to laryngeal vestibule closure, assessed during videofluoroscopic (VF) recording of radio-opaque bolus deglutition.
Modification of brain physiology response to sensory input: | up to 20 min after ingredient ingestion
  Amplitude and latency of the 4 peaks of the pharyngeal sensory evoked potentials (PSEP) on EEG.
Tolerability to the products (gastrointestinal comfort) using a questionnaire, assessed during EEG sessions (V3 and V4) to avoid capturing side effects of the contrast agent (as nausea). | ponctually at the end of visits V3 and V4, after the EEG recording lasting about 30 min, during wich the product is ingested
  using questionnaire
palatability using a questionnaire, assessed during EEG sessions (V3 and V4) | ponctually at the end of visits V3 and V4, after the EEG recording lasting about 30 min, during wich the product is ingested
  using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, Md/PhD, Principal Investigator — Hospital de Mataro
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain